CLINICAL TRIAL: NCT06145581
Title: Remote Monitoring With Health-Coaching for Lifestyle Changes in Older Patients With Multiple Myeloma
Brief Title: Remote Monitoring With Health-Coaching to Improve Quality of Life in Older Patients With Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-005783; NCI-2023-07110 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-005783 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Palliative Care; Interviews as Topic; Remote Patient Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (home-based physical activity) (Experimental): Patients participate in remote monitored home-based physical activity sessions including flexibility practice, slow walking and breathing exercises daily on 6 out of 7 days a week and receive telephone health coaching over 5-20 minutes once a week for 12 weeks. Patients also participate in a brief telephone interview at the end of 12 weeks. Additionally, patients wear a monitor on the wrist to monitor physical activity for 7 days during enrollment and at 3 months.
  Interventions: Behavioral: Supportive Care (home-based physical activity); Other: Exercise Intervention; Other: telephone interview; Other: Remote Monitoring; Procedure: Patient Monitoring; Other: Questionnaire Administration; Other: Electronic Health Record Review

INTERVENTIONS:
Behavioral: Supportive Care (home-based physical activity) — Receive health coaching
Other: Exercise Intervention — Participate in home-based physical activity
Other: telephone interview — Participate in a telephone interview
Other: Remote Monitoring — Undergo remote monitoring
Procedure: Patient Monitoring — Monitor physical activity
Other: Questionnaire Administration — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
This clinical trial tests the effectiveness of a home-based mindfulness physical activity program with remote monitoring combined with structured telephone-based health coaching to decrease fatigue and improve quality of life in older patients with multiple myeloma (MM). Studies have shown that MM patients have the highest symptom burden among all blood cancers, with older patients experiencing more symptoms and problems, such as fatigue and decreased quality of life, compared to younger patients. There is some data to support that physical activity may have beneficial effects on fatigue, physical function, and quality of life in older cancer patients. Studies have also shown that older patients prefer activities that are gentle, holistic, and home-based. Mindfulness-based interventions have been shown to have positive effects on sleep, depression, anxiety and cancer-related fatigue. Health coaching is a patient centered behavioral change intervention that is delivered by various healthcare professionals and involves goal-setting, self-discovery, and accountability. Health coaching interventions have been shown to increase physical activity levels and improve quality of life. A home-based mindfulness physical activity program with remote monitoring combined with structured telephone-based health coaching may decrease fatigue and improve the quality of life in older patients with MM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the effect-size of a novel combined home-based mindfulness physical activity program with telephonic health coaching on 1) patient-reported fatigue assessed by the Brief Fatigue Inventory (BFI) and Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaires and 2) Health-related quality of life assessed by the Patient-Reported Outcomes Measurement Information System Global-10 (PROMIS Global-10) questionnaire, and 3) physical activity levels measured by steps per day.

OUTLINE:

Patients participate in remote monitored home-based physical activity sessions including flexibility practice, slow walking and breathing exercises daily on 6 out of 7 days a week and receive telephone health coaching over 5-20 minutes once a week for 12 weeks. Patients also participate in a brief telephone interview at the end of 12 weeks. Additionally, patients wear a monitor on the wrist to monitor physical activity for 7 days during enrollment and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MM and has received treatment with >= 1 prior lines of treatment, and currently on maintenance treatment with a proteasome inhibitor and/or immunomodulatory agent, and/or anti-C38 antibody
* The ability to read and respond to questions in English
* Age ≥ 65 years
* Moderate or higher fatigue ( > 4) on a scale of 0-10 based on fatigue rating to question: - Rate your average fatigue over the last week, where 0 is no fatigue and 10 is extreme fatigue
* Have wi-fi connection, as the program requires wi-fi to operate

Exclusion Criteria:

* Does not meet listed inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in fatigue - BFI | Baseline; 3 months
  Changes in fatigue will be assessed the Brief Fatigue Inventory (BFI), a 4-item questionnaire asking the participant about their experiences in the past 24 hours. Respondents rate each item from 0 (no fatigue) to 10 (fatigue as bad as you can imagine).
Changes in fatigue - FACIT-F | Baseline; 3 months
  Changes in fatigue will be assessed using the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F). The FACIT-F questionnaire consists of 40 statements designed to assess self-reported fatigue and its impact upon daily activities and function over the past 7 days. Each statement rated on a five-point scale from 0 (not at all) to 4 (very much).

SECONDARY OUTCOMES:
Changes in quality of life - PROMIS-10 | Baseline; 3 months
  The Patient Reported Outcomes Measurement Information System (PROMIS) Global Health questionnaire is a 10-item questionnaire that assess quality of life. All questions have a five-point Likert-type scale, except for the rating of pain which has a ten-point scale.
Effectiveness - qualitative interview | 3 months
  At the end of the 12-week intervention, a member of the study team trained in qualitative interviewing will contact the participant and conduct an interview exploring items such as what the participant found helpful, what improvements they would like, and would they recommend this program to others. The call will be recorded so that it can be transcribed later looking for themes. At the end of the study the recordings will be destroyed.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine H. Abdallah, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials